CLINICAL TRIAL: NCT05446376
Title: Contribution of PET/CT With Gallium 68 Citrate (68Ga-PET/CT) for the Diagnosis of Prosthetic Valve Infective Endocarditis
Acronym: CiGal-EI-TEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/49
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Infective Endocarditis
Keywords: prosthetic valve; PET/CT; Gallium 68; diagnosis; infective endocarditis
MeSH Terms: conditions — Endocarditis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-citrate PET/CT (Experimental)
  Interventions: Drug: 68Ga-citrate PET/CT

INTERVENTIONS:
Drug: 68Ga-citrate PET/CT — PET/CT Imaging with 68Ga-citrate PET/CT injection

SUMMARY:
CiGal-EI-TEP is an exploratory study that aim to assess the diagnostic performance of 68Ga Positron emission tomography (PET) / Computed Tomography (CT) for the diagnosis of prosthetic valve infective endocarditis in comparison with the final diagnosis established according to the ESC 2023 criteria, after 3 months of follow-up, by a panel of experts.

DETAILED DESCRIPTION:
Diagnosis of prosthetic valve infective endocarditis is challenging. It is based on the modified criteria of the European Society of Cardiology (ESC) 2023 which include clinical, microbiological and imaging data. 18F-fluorodeoxyglucose (18FDG) PET/CT is a major diagnostic criterion for prosthetic valve infective endocarditis. In practice, 18FGD-PET/CT is carried out as soon as possible in all patients having valve repair materials and suspected of infective endocarditis on material. According to studies, the sensitivity of 18FDG-PET/CT is around 80% for the diagnosis of infective endocarditis on a prosthetic valve. The use of 18FDG requires a low carbohydrate diet the day before the exam. Compliance with this condition is difficult to obtain, in diabetic patients. Without following these instructions, interpretation of the heart valves is difficult, and this can leed to false negatives. The use of an another radiopharmaceutical drug could avoid these problem. PET/CT with Gallium 68 citrate (68Ga-PET/CT) could reduce the number of false negatives while having similar specificity to 18FDG-PET/CT for the diagnosis of infective endocarditis on prosthetic valve.

The investigators therefore propose an exploratory study to assess the diagnostic performance of 68Ga-PET/CT for the diagnosis of prosthetic valve infective endocarditis in comparison with the final diagnosis established according to the ESC 2023 criteria, after 3 months of follow-up, by a panel of experts.

Patient suspected of infective endocarditis on prosthetic valves will be included.

The index test (68Ga-PET/CT) and the usual test (18FDG-PET/CT) will be performed in all participants. The 68Ga-PET/CT will be performed the day before, the same day or the next day after 18FDG-PET/CT.

. Both PET/CT scans will be interpreted independently by two experienced nuclear physicians, blinded to the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (over 18 years old);
* patient with a prosthetic heart valve;
* patient suspected of infective endocarditis (on clinical and/or microbiological and/or imaging data);
* patient whose history is discussed in the multidisciplinary meeting dedicated to endocarditis;
* patient beneficiary of a social security scheme;
* free, informed and written consent signed by the participant and the investigator.

Exclusion Criteria:

* pregnant or breastfeeding women;
* women of childbearing potential not using effective contraception;
* patients referred to in articles L.1121-5 to L.1121-8 (persons deprived of liberty by judicial or administrative decision, minors, adults subject to a legal protection measure or unable to express their consent);
* subject in a period of relative exclusion due to another protocol;
* known contraindication to PET/CT with injection of radiotracers (hypersensitivity to radiopharmaceuticals and/or excipients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-PET/CT for the diagnosis of prosthetic valve infective endocarditis in patients suspected of infective endocarditis on prosthetic valve | 3 months after baseline (Day 0)
  The final diagnosis of infective endocarditis is established according to the ESC 2023 criteria (assessed at 3 months by a panel of experts).

SECONDARY OUTCOMES:
Diagnostic accuracy of 68Ga citrate PET / CT scan CT for prosthetic valve infective endocarditis in patients suspected of infective endocarditis on prosthetic valve | 3 months after baseline (Day 0)
  Specificity, positive and negative predictive values of 68Ga-PET/CT for the diagnosis of infective endocarditis on prosthetic valve in patients suspected of infective endocarditis on prosthetic valve.
Inter-observer reproducibility of 68Ga-citrate PET/CT interpretation | 3 months after baseline (Day 0)
  Intraclass correlation coefficient and/or Cohen's Kappa.
Comparison of diagnostic accuracy of 68Ga-PET/CT and 18FDG-PET/CT for the diagnosis of infective endocarditis on prosthetic valve. | 3 months after baseline (Day 0)
  Sensitivity, specificity and positive and negative predictive values of 18FDG-PET/CT for the diagnosis of infective endocarditis on prosthetic valve.
o Agreement between 68Ga-PET/CT and 18FDG-PET/CT for the evaluation of the spread of infection assessment and the search for the initial portal of pathogen entry | 3 months after baseline (Day 0)
  Cohen's Kappa

CONTACTS AND LOCATIONS:
Overall Officials: Carine GREIB, MD, Principal Investigator — University Hospital, Bordeaux; Eric FRISON, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No